CLINICAL TRIAL: NCT05690048
Title: Fecal Microbiota Transfer in Liver Cancer to Overcome Resistance to Atezolizumab/Bevacizumab (FLORA)
Acronym: FLORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Dill (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other); German Cancer Research Center (Other); Heidelberg University (Other); University of Cologne (Other); Universitätsmedizin Mannheim (Other)
Responsible Party: Sponsor-Investigator, Michael Dill, Principal Investigator, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Version 3.1/11.02.2025
Record Dates: First submitted 2022-12-13; First posted 2023-01-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Immunotherapy; HCC - Hepatocellular Carcinoma
Keywords: immunotherapy; fecal microbiota transfer; HCC; gut microbiota; tumor microenvironment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fecal Microbiota Transplantation; Vancomycin; atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, placebo-controlled, double-blind, phase II with two arms (verum/placebo) in a parallel group design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin + A/B + FMT (Experimental): 1. Atezolizumab 1200mg i.v. & Bevacizumab 15mg/kg body weight i.v. (A/B) as standard of care (SOC).
  2. Vancomycin orally (250 mg 4xd, day -3 to 0) for reduction of original patient gut microbiota.
  3. Fecal microbiota transfer (FMT) via capsules (total 50 g of fecal matter) on day 0 and day 21.
  Interventions: Drug: Fecal microbiota transfer; Drug: Vancomycin Oral Capsule; Drug: Atezolizumab + Bevacizumab
- Placebo Vancomycin + A/B + Placebo FMT (Placebo Comparator): 1. Atezolizumab 1200mg i.v. & bevacizumab 15mg/kg body weight i.v. (A/B) as standard of care (SOC).
  2. Placebo vancomycin orally (4xd, day -3 to 0) for reduction of original patient gut microbiota.
  3. Placebo fecal microbiota transfer (FMT) via capsules on day 0 and day 21.
  Interventions: Drug: Atezolizumab + Bevacizumab; Drug: Placebo Vancomycin Oral Capsule; Drug: Placebo Fecal microbiota transfer

INTERVENTIONS:
Drug: Fecal microbiota transfer — FMT via capsule (50 g of fecal matter) on day 0 and day 21.
  Other Names: FMT; INTESTIFIX 001
  Arms: Vancomycin + A/B + FMT
Drug: Vancomycin Oral Capsule — Vancomycin orally (250 mg 4xd, day -3 to 0).
  Arms: Vancomycin + A/B + FMT
Drug: Atezolizumab + Bevacizumab — Atezolizumab 1200mg i.v. & Bevacizumab 15mg/kg body weight i.v. (A/B) as standard of care (SOC).
  Other Names: A/B
Drug: Placebo Vancomycin Oral Capsule — Placebo Vancomycin orally (4xd, day -3 to 0).
  Arms: Placebo Vancomycin + A/B + Placebo FMT
Drug: Placebo Fecal microbiota transfer — Placebo Fecal microbiota transfer (FMT) via capsule on day 0 and day 21.
  Other Names: Placebo FMT; Placebo INTESTIFIX 001
  Arms: Placebo Vancomycin + A/B + Placebo FMT

SUMMARY:
The interventional, randomized, placebo-controlled, double-blind phase II-trial FLORA will assess safety and immunogenicity of fecal microbiota transfer in combination with standard of care immunotherapy in advanced hepatocellular carcinoma (HCC) in a parallel group design.

Subjects will be randomized 2:1 into either the FMT or placebo group.

DETAILED DESCRIPTION:
Eligible HCC patients visiting the outpatient clinics at the study sites of the NCT Germany will be enrolled into the study after informed consent. Patients undergo 2:1 randomization into either the FMT or placebo group. Prior to the intervention, a sigmoidoscopy with mucosal biopsies will be performed. At day -3 to 0 oral Vancomycin 4x 250mg or placebo will be given. Atezolizumab/bevacizumab (A/B) will be administered as standard of care every 21 days, starting on day 0. At day 0 and 21, concurrent to the first and second cycle of A/B, encapsulated FMT or placebo will be administered on the same day. At day 40-42, before the third cycle of A/B, a tumor biopsy and a sigmoidoscopy will be performed. The first radiologic assessment will be performed after 4 cycles of A/B. Clinical efficacy and safety will be assessed as indicated per protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Confirmed radiologic or histological diagnosis of HCC
3. Disease not amenable to resection, liver transplantation or loco-regionary therapy
4. Eligible for therapy with Atezolizumab / Bevacizumab according to standard of care
5. Measurable disease per RECIST 1.1
6. Preserved liver function with a Child-Pugh score A or B (maximally 7 points)
7. Performance status ECOG 0-1

Exclusion Criteria:

1. Use of immunosuppressive medication within 6 months prior to the first dose of Atezolizumab / Bevacizumab.
2. Active or prior documented autoimmune or inflammatory disorders
3. Prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-VEGF antibodies.
4. Known to have tested positive for human immunodeficiency virus (HIV) infection.
5. Co-infection of HBV and HCV. Subjects with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV.
6. Evidence by investigator assessment of varices at risk of bleeding on upper endoscopy undertaken within 12 months of randomization.
7. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow a formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism or excretion of investigational product.
8. Uncontrolled arterial hypertension defined by a systolic pressure > 150 mm Hg or diastolic pressure > 90 mm Hg or other hypertensive cardiovascular complications despite standard medical treatment.
9. Any history of nephrotic or nephritic syndrome.
10. Usage of systemic antibiotic therapy within 2 weeks prior to the first dose of Atezolizumab/Bevacizumab.
11. Usage of probiotic products/supplements within 1 week prior to the first dose of Atezolizumab/Bevacizumab.
12. Known fibrolamellar HCC, sarcomatoid HCC, infiltrative-type HCC, or mixed cholangiocarcinoma and HCC.
13. History of another primary malignancy.
14. Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention.
15. Pregnancy or lactation.
16. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
17. Participation in other interventional clinical trials or observation period of competing clinical trials, respectively.
18. Held in an institution by legal or official order.
19. Legally incapacitated.
20. Known hypersensitivity to any component of the vancomycin, atezolizumab or bevacizumab formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of immunogenicity | 6 weeks after treatment initiation
  Tumoral CD8+ T cell infiltration after 2 cycles of treatment with Vancomycin, A/B + FMT in comparison to Vancomycin-placebo, A/B + FMT-placebo
Safety of the therapeutic combination in advanced HCC | The observational period begins with the first administration of the 1st IMP (Vancomycin/Placebo) on day -3 and ends with either the Follow-up visit after 15 weeks (Day 105) or the initiation of a subsequent anticancer treatment.
  Occurence of Adverse Events (AE) & immune-related adverse events (irAE)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment until the date of death from any cause, assessed up to 4 years.
  To evaluate the efficacy of Vancomycin, A/B + INTESTIFIX 001 in comparison to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Overall Survival (OS).
  OS is defined as the time from start of treatment (first dose of A/B) to time of death from any cause in days. Administrative censoring is applied for patients who survive the end of the trial. Death cases will either become known during the clinical study treatment, or information will be obtained on the occasion of follow-up calls, or from e.g. treating physicians. Otherwise, patients for whom the date of death is unknown are censored at the last time point they are known to be alive.
Progression free survival (PFS) | From start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years.
  To evaluate the efficacy of Vancomycin, A/B + INTESTIFIX 001as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Progression Free Survival (PFS).
  PFS is defined as the time from start of treatment (first dose A/B) until objective tumor progression as determined by the radiologist per RECIST 1.1 or death, whichever occurs first.
Disease control (DC) | From start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years.
  To evaluate the efficacy of Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Disease Control (DC). DC is defined as achieving complete response (CR), partial response (PR) or stable disease (SD) as best overall response during observation period as determined by the radiologist per RECIST 1.1 criteria.
Objective Response (OR) | From start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years.
  To evaluate the efficacy of Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Objective Response (OR).
  OR is defined as tumor size reduction, meaning PR or CR, as determined by the radiologist per RECIST 1.1 criteria assessed by best overall response during the observation period.
Duration of Response (DoR) | From start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years.
  To evaluate the efficacy of Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Duration of Response (DoR).
  DoR is defined as the time from first documented response (either PR or CR per RECIST 1.1, whichever is recorded first) to first subsequent progression (first assessment of PD per RECIST 1.1 or death). DoR is only defined for the patients who experienced a response.
AFP serological response rate | From start until end of treatment (11 weeks).
  To evaluate the efficacy Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to AFP serological response rate.
  AFP serological response rate is defined as defined as a >20% de- crease in serum AFP (ng/ml)
Hepatic Function measured by model of end-stage liver disease (MELD) score | From start until end of treatment (11 weeks).
  To evaluate the efficacy Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Hepatic function measured by model of end-stage liver disease (MELD) score (Range 6-40 points, with higher points indicating worsening of function).
  The hepatic function endpoints are the absolute scores at all assessed time points as well as the change to baseline.
Hepatic Function measured by Child-Pugh score | From start until end of treatment (11 weeks).
  To evaluate the efficacy Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Hepatic function measured by Child-Pugh Score (CPS) (Range 5-15, with higher scores indicating worsening).
  The CPS endpoints are the absolute scores at all assessed time points as well as the change to baseline.
Hepatic Function measured by ALBI grade | From start until end of treatment (11 weeks).
  To evaluate the efficacy Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Hepatic function measured by ALBI grade (Range 1-3, with higher scores indicating worsening).
  The ALBI grade endpoints are the absolute scores at all assessed time points as well as the change to baseline.
Hepatic Function measured by Psychometric Hepatic Encephalopathy Score (PHES) | From start until end of treatment (11 weeks).
  To evaluate the efficacy Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo with respect to Hepatic function measured Psychometric Hepatic Encephalopathy Score (PHES) questionnaire (Range -15 tp +15, with higher scores indicating better cognitive function).
  The PHES endpoints are the absolute scores at all assessed time points as well as the change to baseline.
Health-related quality of life - general | From start until end of treatment (11 weeks).
  To evaluate the effect of Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo in respect to Health-related quality of life. Patient reported outcomes (PRO) via are assessed by questionnaire (EORTC QLQ-C30) and are collected during treatment. Final scores are transformed such that they range from 0 to 100, where higher scores indicate greater level of symptoms. The PRO endpoints are the absolute scores at all assessed time points as well as the change to baseline.
Health-related quality of life - disease-specific | From start until end of treatment (11 weeks).
  To evaluate the effect of Vancomycin, A/B + INTESTIFIX 001 as relative to Vancomycin-placebo, A/B + INTESTIFIX 001-placebo in respect to Health-related quality of life. Patient reported outcomes (PRO) are assessed by HCC-specific questionnaire (EORTC QLQ-HCC18) and are collected during treatment. Final scores are transformed such that they range from 0 to 100, where higher scores indicate greater level of symptoms. The PRO endpoints are the absolute scores at all assessed time points as well as the change to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Dill, PhD, Principal Investigator — University Hospital Heidelberg, Heidelberg, Baden-Württemberg 69120
Locations (7):
- Germany (7):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Hospital Augsburg, Augsburg
  - University Hospital Essen, Essen
  - University Hospital Mannheim, Mannheim
  - University Hospital Regensburg, Regensburg
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Rauber C, Roberti MP, Vehreschild MJ, Tsakmaklis A, Springfeld C, Teufel A, Ettrich T, Jochheim L, Kandulski A, Missios P, Mohr R, Reichart A, Waldschmidt DT, Sauer LD, Sander A, Schirmacher P, Jager D, Michl P, Dill MT. Protocol: Faecal microbiota transfer in liver cancer to overcome resistance to atezolizumab/bevacizumab - a multicentre, randomised, placebo-controlled, double-blind phase II trial (the FLORA trial). BMJ Open. 2025 Sep 9;15(9):e097802. doi: 10.1136/bmjopen-2024-097802. PMID 40930564